CLINICAL TRIAL: NCT04354961
Title: Aumolertinib as First-line Treatment in EGFR-Mutant Pulmonary Adenosquamous Carcinoma: A Multicenter, Single-Arm, Prospective Study (ARISE)
Brief Title: Almonertinib as First-line Treatment in Patients With EGFR+ Positive Pulmonary Adenosquamous Carcinoma or Combined Adenocarcinoma and Squamous Cell Carcinoma
Acronym: ARISE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-LK-2020-003
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Adenosquamous Carcinoma
MeSH Terms: interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Almonertinib 110mg PO once daily (Experimental)
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — Almonertinib 110mg PO once daily. A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Investigational Product

SUMMARY:
This is a prospective, multi-center, single-arm clinical trial.

DETAILED DESCRIPTION:
This is a multicenter, single arm, phase II study assessing the efficacy and safety of Almonertinib as first-line treatment in patients with EGFR mutation positive locally advanced or metastatic Pulmonary Adenosquamous Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures, sampling and analyses.
* Male or female, age at least 18 years.
* Pathologically confirmed locally advanced or metastatic pulmonary adenosquamous carcinoma. Patients must be treatment-naïve for locally advanced or metastatic pulmonary adenosquamous carcinoma. provided all other entry criteria are satisfied.
* Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) if 6 months or more have passed since completion of therapy.
* The tumour harbours EGFR genes mutations assessed by central testing using tissue, blood, pleural effusion, peritoneal effusion, and cerebrospinal fluid samples..
* A WHO performance status equal to 0-2 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements. If only one measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and baseline tumour assessment scans are done at least 14days afar the screening biopsy is performed.
* Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at Screening:

  1. Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
  2. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.
  3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
* Male patients should be willing to use barrier contraception (i.e., condoms).
* For inclusion in study, patient must provide a written informed consent.

Exclusion Criteria:

* Treatment with any of the following:

  1. Prior treatment with an EGFR TKI.
  2. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
  3. Radiotherapy with a limited field of radiation for palliation within 4 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
  4. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug.
* Patients with other malignancies requiring standard treatment or major surgery within 2 years after the first dose of study treatment, except basal cell carcinoma and carcinoma in situ.
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection. Screening for chronic conditions is not required.
* Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of Almonertinib.
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTc) > 470 ms obtained from electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
  2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
  4. Left ventricular ejection fraction (LVEF) ≤ 40%.
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

  1. Absolute neutrophil count (ANC) <1.5×109 / L
  2. Platelet count <100×109 / L
  3. Hemoglobin <90 g/L（<9 g/dL）
  4. Alanine aminotransferase > 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
  5. Aspartate aminotransferase (AST) > 2.5 × ULN if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
  6. Total bilirubin (TBL) > 1.5 × ULN if no liver metastases or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
  7. Creatinine > 1.5 × ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 × ULN.
* Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.
* History of hypersensitivity to any active or inactive ingredient of Almonertinib or to drugs with a similar chemical structure or class to Almonertinib.
* Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
* Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
* Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From baseline, then every 6 weeks, until disease progression or discontinuation from study. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  To assess the efficacy of Almonertinib as first line therapy to EGFRm+, locally advanced or metastatic Pulmonary Adenosquamous Carcinoma patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Assess the anti-tumor activity: OS | Start of study drug to Survival Endpoint through study completion, an average of 4 years.
  Overall survival (OS)
Assess the anti-tumor activity: ORR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression assessed up to 24 months.
  Objective response rate (ORR)
Assess the anti-tumor activity: DCR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. The DCR is defined as the proportion of patients with a best overall response of CR, PR, or SD assessed up to 24 months.
  Disease control rate (DCR)
Assess the anti-tumor activity: DoR | DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression assessed up to 24 months.
  Duration of response (DoR)
Assess the safety of Almonertinib : Number of AEs/SAEs | Continuously throughout the study until 28 days after Termination of the treatment
  Number of adverse events (AEs)/serious adverse events (SAEs)
QoL QoL | 2 years
  To assess disease-related symptoms and QoL in overall population as well as in pre-specified subgroups
Assess the anti-tumor activity: iORR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression assessed up to 24 months.
  Intracranial Objective response rate (iORR)
Assess the anti-tumor activity: iDCR | From baseline, then every 6 weeks, until disease progression or discontinuation from study. ORR is defined as the percentage of patients who have at least 1 response of CR or PR prior to any evidence of progression assessed up to 24 months.
  Intracranial Disease control rate (iDCR)
Intracranial Progression Free Survival (iPFS) | From baseline, then every 6 weeks, until disease progression or discontinuation from study. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  To assess the efficacy of Almonertinib as first line therapy to EGFRm+, locally advanced or metastatic Pulmonary Adenosquamous Carcinoma patients by assessment of intracranial progression free survival (iPFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Hunan Cancer Hospital, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xinqiao Hospital, Army Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Provincial Hospital, Fuzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - The second Affiliated Hospital of Kunming Medical University, Kunming
  - The second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tongji Hospital of Tongji Medical College,Huazhong University of Science and Technology, Wuhan
  - Air Force Medical University of PLA (the Fourth Military Medical University), Xi'an
  - Henan Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No